CLINICAL TRIAL: NCT00573924
Title: Prospective Randomized Comparison of the Effect of Frequent Oral Dosing Versus Constant IV Infusion of Proton Pump Inhibitor on Intragastric pH in Patients With Bleeding Ulcers
Brief Title: Trial of Oral Versus Intravenous Proton Pump Inhibitor on Intragastric pH in Patients With Bleeding Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Loren Laine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-06-00014; HS-06-00014
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Peptic Ulcer Hemorrhage
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Proton Pump Inhibitors; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Oral PPI
  Interventions: Drug: Proton pump inhibitor (lansoprazole)
- 2 (Active Comparator): Intravenous PPI
  Interventions: Drug: Proton pump inhibitor (lansoprazole)

INTERVENTIONS:
Drug: Proton pump inhibitor (lansoprazole) — 1. 120 mg PO and then 30 mg PO q 3 h from 3 to 21 hrs
  2. 90 mg IV bolus followed 9 mg/hr infusion for 24 hrs

SUMMARY:
Patients with bleeding ulcers identified by endoscopy will be randomly assigned to receive an acid-blocking drug (called a proton pump inhibitor [PPI]) either by mouth every 3 hours for 24 hours or intravenously (IV) by constant infusion for 24 hours. A pH probe in the stomach will be used to determine intragastric pH (a measure of the acid production in the stomach) at baseline and during the 24 hours of therapy. The purpose of the study is to determine if the continuous intravenous administration of the drug provides better reduction of acid in the stomach than the oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to hospital with overt upper GI bleeding and found to have an ulcer as the cause on endoscopy

Exclusion Criteria:

* Previous gastric surgery
* Active bleeding at end of endoscopy (despite hemostatic therapy)
* Recent PPI or H2RA use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-02; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Intragastric pH > 6 | 24 hours

SECONDARY OUTCOMES:
Mean intragastric pH | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Loren Laine, M.D., Principal Investigator — University of Southern California
Locations (1):
- L.A. County + U.S.C. Medical Center, Los Angeles, California, United States

REFERENCES:
- [Result] Laine L, Shah A, Bemanian S. Intragastric pH with oral vs intravenous bolus plus infusion proton-pump inhibitor therapy in patients with bleeding ulcers. Gastroenterology. 2008 Jun;134(7):1836-41. doi: 10.1053/j.gastro.2008.03.006. Epub 2008 Mar 10. PMID 18423628